CLINICAL TRIAL: NCT04778553
Title: Clinical Evaluation of the iMOST Analyzer - Matrix Study Comparing Capillary and Venous Whole Blood
Brief Title: Clinical Evaluation of the iMOST-X1 Hematology Analyzer - Matrix Study
Status: Completed | Type: Observational
Sponsor: Essenlix Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: ESX-iMOST-X1-3
Record Dates: First submitted 2021-02-26; First posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Hematologic Tests
Keywords: CBC, WBC, Hemoglobin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: iMOST X-1 Hematology Analyzer — The X-1 is a point of care automated hematology analyzer

SUMMARY:
This is a method comparison study for an in vitro diagnostic device. The device is a point of care automated hematology analyzer which measures CBC parameters with a small drop of venous or capillary, e.g., fingerstick blood. The study compared the CBC results from the test device, the Essenlix iMOST X-1 to the predicate laboratory based Horiba Pentra 60C+ analyzer. The CBC parameters were hemoglobin, White Blood Cells (WBC) and the WBC Differential for Granulocytes, Neutrophils, Lymphocytes and Monocytes. The study subjects were patient donors (age 18 and older) attending the hospital clinic from whom Informed Consent had been received.

DETAILED DESCRIPTION:
These studies demonstrate that the iMOST X-1 system yields equivalent results to the Horiba predicate system when using either capillary and venous blood specimens. Furthermore, there are three alternative methods of capillary blood sampling for the iMOST and all have direct applicability to the iMOST system. As has been published in the peer reviewed literature, different fingerstick sample collection methods yield slightly different CBC results, specifically the WBC and the WBC Differential. The iMOST employs an integrated software algorithm with which the use can employ site specific calibration constants to correctly match the selected capillary blood specimen to the venous specimen for the WBC test results. All three methods of blood collection are thus described in the "Instructions for Use".

ELIGIBILITY:
Inclusion Criteria:

* all clinic attendees

Exclusion Criteria:

* unable to provide a venous and fingerstick blood specimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients attending the hospital outpatient clinic who had voluntarily consented to blood donation for venous and capillary blood collection
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2020-12-09 (Actual); Study Completion 2021-01-21 (Actual)

PRIMARY OUTCOMES:
Method Comparison of CBC Results | October- December 2020
  Blood Diagnostic Tests for CBC

CONTACTS AND LOCATIONS:
Overall Officials: Megha Shah, M.D., Principal Investigator — Hunterdon Medical Center
Locations (1):
- Hunterdon Medical Center, Flemington, New Jersey, United States